CLINICAL TRIAL: NCT07345273
Title: Reporting of Tumour Deposits in Colorectal Cancer by Radiology and Pathology
Acronym: RADAR
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Croydon Health Services NHS Trust (Other); Epsom and St Helier University Hospitals NHS Trust (Other); Basingstoke and North Hampshire Hospital (Unknown); London North West University Health Care NHS Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 183491
Record Dates: First submitted 2025-12-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Rectal Adenocarcinoma
Keywords: Rectal Adenocarcinoma; Tumour Deposits; TNM staging; Extramural Venous Invasion
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TNM5: Patients with rectal cancer diagnosed between 2007-2017 who were staged using TNM5
  Interventions: Other: No Intervention: Observational Cohort
- TNM8: Patients with rectal cancer diagnosed between 2022-2024 who were staged using TNM8
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention is to be performed. This is an observational retrospective cohort study only

SUMMARY:
Recent research shows that tumour deposits-small spots of cancer found near the main bowel tumour-may give doctors important information about how aggressive the cancer is and how likely it is to come back.

Doctors can find tumour deposits either:

1. When looking at scans before surgery, or
2. when examining the removed bowel tissue under the microscope after surgery.

In the past, tumour deposits were not always recorded properly. This is because older cancer-staging systems (called TNM 5) used in the UK treated these spots differently, depending on their size, and sometimes labelled them as lymph nodes even when they were not. As a result, many tumour deposits were missed in reports.

Since 2018, the UK has been using an updated staging system (called TNM 8) that gives tumour deposits their own category. This means doctors are now expected to report them separately when they are found in the tissue around the bowel.

This matters because the investigators know that patients who have tumour deposits may have a higher risk of the cancer returning or spreading. Because of this, these patients might benefit from extra treatment-such as chemotherapy or radiotherapy-on top of surgery.

However, if tumour deposits are not routinely recorded on scans or pathology reports, doctors may not realise a patient has them. This means that:

1. Patients may not get the most appropriate advice about their cancer, and
2. Patients may miss out on treatments that could help reduce the chance of the cancer returning.

This research project aims to find out two things:

1. Are tumour deposits being routinely reported on scans and pathology reports for rectal cancer since the newer TNM 8 system was introduced? And
2. Is there a link between reporting tumour deposits and another important finding called EMVI (extramural vascular invasion), which also affects cancer behaviour and treatment decisions?

DETAILED DESCRIPTION:
Background:

There is increasing evidence that Tumour Deposits (TDs) play an important role in determining prognosis in colorectal cancer patients, both on pathology and on pre-operative imaging (1-2). There is a great variation in their reported prevalence on pathology (1) depending on the staging system and pathology techniques used. Previous work to determine the prevalence of TDs in the UK has relied on the TNM 5 classification, since the 6th and 7th editions were not adopted into UK practice. In TNM 5, all tumour nodules of >3mm were classified as lymph nodes, regardless of whether there was evidence of underlying nodal architecture. Nodules of under 3mm were included in the T stage. Reporting of TDs only took place if the pathologist made specific mention of them in the body of the report, therefore the reported prevalence was very low (6%) compared to when detected on imaging (36%)(2). TNM 8, released in 2017, is the current Tumour Node Metastases staging system used for colorectal cancer (3) and was adopted in the UK from January 2018 onwards. In TNM 8 however, TDs in the subserosa, or in non-peritonealised pericolic or perirectal soft tissue without regional lymph node metastatic disease are reported as N1c. The aim of this multicentre retrospective evaluation is to understand if TDs are being routinely reported in imaging and pathology in rectal cancer patients since the introduction of TNM 8.

Rationale:

There is increasing evidence that TDs impact the recurrence of cancer and cancer death in patients with rectal cancer for the worse. These patients may therefore benefit from additional treatment with chemotherapy or radiotherapy. However, if we are not recording TDs routinely, and don't know at the time of deciding how to treat these patients that they have TDs, then we are not counselling patients properly as well as may not be offering them additional chemotherapy or radiotherapy.

Objectives:

Primary Objectives:

To determine whether, since the introduction of TNM 8, TDs are being routinely reported in staging of rectal cancer on imaging and pathology

Secondary Objective:

To determine if there is as positive association between the reporting of TDs and the reporting of Extramural Venous Invasion.

References:

Please see separate References Section

ELIGIBILITY:
Inclusion Criteria:

1. Primary adenocarcinoma of the rectum (proven by biopsy)
2. Undergone surgical resection between 01st January 2007 to 31st December 2017 inclusive for the TNM 5 cohort
3. Undergone surgical resection between 01st January 2022 to 31st December 2024 inclusive for the TNM 8 cohort

3. Staging with MRI reports are available 4. Post-operative pathology report available 5. Patients aged 16 years and over

Exclusion Criteria:

1. Synchronous metastatic tumours
2. Under the age of 16 years
3. MRI and/or pathology reports are not available

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (>16 years old) with primary adenocarcinoma of the rectum who have undergone resectional surgery
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of Tumour Deposits | For MRI: MRI reporting within 8 weeks prior to surgery For pathology: Pathology reporting up to 4 weeks after surgery
  1. The frequency of Tumour Deposits on MRI in the TNM 8 cohort compared to TNM 5 cohort and
  2. The frequency of Tumour Deposits on pathology in the TNM 8 cohort compared to TNM 5 cohort

SECONDARY OUTCOMES:
The correlation between reporting of tumour deposits and extramural venous invasion | For MRI: MRI reporting within 8 weeks prior to surgery For pathology: Pathology reporting up to 4 weeks after surgery
  1. The percentage of patients with extramural venous invasion on MRI among patients with MRI-detected tumour deposits. Measurement tool is standardised colorectal cancer pelvic MRI reporting.
  2. The percentage of patients with histopathological extramural venous invasion among patients with histopathologically confirmed tumour deposits. Measurement tool is standardised colorectal cancer histopathology reporting.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Croydon Health Services NHS Trusts, Croydon, Select Your County
  - London North West University Healthcare NHS Trust, London, Select Your County
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Epsom and St Helier University Hospitals NHS Trust, Surrey Quays

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared. At the time of publication of results, fully anonymised data will be made available to those that request it upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol which includes the statistical analysis plan is available for sharing immediately. Results will be available at the time of publication.
Access Criteria: Anyone will be able to access the IPD and supporting information. The will be able to access the study protocol which includes the statistical analysis plan and anonymised individual participant data. They can access it by emailing Prof. Brown or Harpreet Sekhon at gina.brown@imperial.ac.uk, giclinicaltrials@imperial.ac.uk or hks224@ic.ac.uk Alternatively, it will be released onto the ClinicalTrials.gov record at the time of Results publication

REFERENCES:
- [Background] Amin MB, Edge SB, Greene FL, et al., editors. AJCC cancer staging manual. 8th ed. New York: Springer; 2017.
- [Background] Sekhon Inderjit Singh HK, Lord A, Pawa N, Brown G. The Prognostic Impact of Imaging Detected Tumor Deposits in Rectal Cancer: A Systematic Review and Meta-analysis. Ann Surg Oncol. 2026 Jan;33(1):199-209. doi: 10.1245/s10434-025-18371-w. Epub 2025 Sep 30. PMID 41028637
- [Background] Lord AC, D'Souza N, Pucher PH, Moran BJ, Abulafi AM, Wotherspoon A, Rasheed S, Brown G. Significance of extranodal tumour deposits in colorectal cancer: A systematic review and meta-analysis. Eur J Cancer. 2017 Sep;82:92-102. doi: 10.1016/j.ejca.2017.05.027. Epub 2017 Jun 23. PMID 28651160